CLINICAL TRIAL: NCT02657421
Title: A Multi-Center, Prospective, Observational Study to Assess Outcomes for Patients Treated for Lumbar Spinal Conditions Using an OLIF25™ and/or OLIF51™Approach
Brief Title: OLIF25™ /OLIF51™ Study
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-05
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2017-07

CONDITIONS: Degenerative Disc Disease; Scoliosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Oblique Lateral Interbody Fusion — The oblique lateral interbody fusion (OLIF) procedures at L2-L5 (OLIF25™) and L5-S1 (OLIF51™) is a minimally invasive surgical option for degenerative lumbar disease. This approach allows for psoas-preserving access to the lumbar spine and minimizes the need to reposition the patient during surgery for accessing additional spinal levels for the interbody fusion portion of the procedure
  Other Names: OLIF

SUMMARY:
The purpose of this single-arm observational study is to observe and document clinical outcomes of the OLIF25™ and OLIF51™ procedures in patients diagnosed with degenerative disc disease or degenerative scoliosis, and report the rate of adverse events of interest through the 24 months follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older.
2. Patient agrees to participate in the study and is able to sign the informed consent/data release form.
3. Patient is undergoing surgery from L2-L5 for OLIF25™ and/or from L5-S1 for OLIF51™ for degenerative disc disease or degenerative scoliosis.

Exclusion Criteria:

1. Illiterate or vulnerable patients (e.g. minors, participants incapable of judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have surgery from L2-L5 for OLIF25™ and/or from L5-S1 for OLIF51™ for degenerative disc disease or degenerative scoliosis.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Back and Leg Pain Measured by Visual Analogue Scales (VAS) | 24 months
Oswestry Disability Index (ODI) | 24 months
European Quality of Life-5 Dimensions (EQ-5D) self-report questionnaire | 24 months
Neurological deficits assessed by neurological status | 24 months
  Neurological status is based on seven components of measurements: Motor function; Sensory function; Deep Tendon reflexes; Sympathetic Exam; Claudication; Urinary bladder retention/Bowel retention; and Sexual Dysfunction.
Rate of adverse events | 24 months

OTHER OUTCOMES:
Surgical Data | Day 0 to Day 5
  Surgical data include mean blood loss, operative time, and length of hospital stay (LOS).
Work status | 24 months
Spino-Pelvic Measurements by X-ray | 24 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Advanced Neurosurgery Associates, Murrieta, California
  - University of California San Francisco (UCSF), San Francisco, California
  - The B.A.C.K. Center, Melbourne, Florida
  - Foundation for Orthopaedic Research and Education (FORE), Tampa, Florida
  - NewYork-Presbyterian/The Allen Hospital, New York, New York
  - Alleghany Health Network Research Institute, Pittsburgh, Pennsylvania
- Ste Elisabeth hospital, Brussels, Belgium
- FN Ostrava, Ostrava, Poruba, Czechia
- Clinique Du Mail, La Rochelle, France
- Azienda Ospedaliera - Ospedale Civile di Legnano, Legnano, Italy
- CUF Descobertas, Lisbon, Portugal
- Orthospine Group, San Juan, Puerto Rico